CLINICAL TRIAL: NCT01642030
Title: Analgesic Effects and Abuse Liability of Intravenous Hydromorphone and Buprenorphine in Pain-free Opioid Dependent Participants
Brief Title: Study of the Treatment of Experimental Pain in Opioid Dependent Persons on Methadone or Buprenorphine Maintenance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00071459; K23DA029609 (NIH); 1203 (Other: PI)
Record Dates: First submitted 2012-07-09; First posted 2012-07-17 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Opioid Dependence; Pain; Addiction
Keywords: Quantitative sensory testing; Cold pressor test; Opioid dependence; Methadone maintenance; Buprenorphine maintenance; Abuse liability; Diffuse Noxious Inhibitory Controls (DNIC); Temporal Summation
MeSH Terms: conditions — Opioid-Related Disorders; Pain; Behavior, Addictive | interventions — Saline Solution; Hydromorphone; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone Maintenance (Other)
  Interventions: Drug: Placebo; Drug: Hydromorphone
- Buprenorphine Maintenance (Other)
  Interventions: Drug: Placebo; Drug: Hydromorphone; Drug: Buprenorphine

INTERVENTIONS:
Drug: Placebo — Intravenous injection of approximately 5 mL administered via slow push over 5 minutes. Given 4 injections during the session with each injection separated by 1.5 hours.
  Other Names: Normal Saline
Drug: Hydromorphone — Intravenous injection of approximately 5 mL administered via slow push over 5 minutes. Given 4 injections during the session with each injection separated by 1.5 hours.
  Other Names: Dilaudid
Drug: Buprenorphine — Intravenous injection of approximately 5 mL administered via slow push over 5 minutes. Given 4 injections during the session with each injection separated by 1.5 hours.
  Other Names: Suboxone; Subutex
  Arms: Buprenorphine Maintenance

SUMMARY:
Pain is very common in persons with a history of addiction, but few studies have examined the best treatment of pain in this population. This is a study to determine the pain relief provided by intravenous hydromorphone (Dilaudid) or buprenorphine given to persons maintained on stable doses of methadone or buprenorphine. Experimental sessions will require overnight stays on a residential research unit. In these sessions, persons will be exposed to standard experimental pain techniques at baseline and then rate the relief (if any) provided by the study medication when exposed to the same techniques. Persons will be asked to participate in 2 or 3 sessions, each separated by at least 7 days.

DETAILED DESCRIPTION:
This research is being done to learn how to better treat pain in people maintained on opioid medications, like methadone and buprenorphine (Suboxone ®, Subutex ®). People who take opioid medications for long periods of time are known to experience pain differently; and, regular amounts of medications may not be enough to treat the pain of these individuals. Additionally, many people with a history of addiction are afraid of taking opioid pain relievers, like morphine or hydromorphone (Dilaudid ®), for fear of relapse.

This study will help guide the medical community on better pain treatment for people prescribed buprenorphine or methadone. Investigators also want to determine the risk for relapse in people who receive opioid pain relievers for the treatment of acute pain.

Healthy people aged 18-55 who are maintained on buprenorphine or methadone for the treatment of opioid dependence may take part in this study. Participants must be free of illicit drug use and be on a stable dose of methadone or buprenorphine. Initial screening will occur over the phone and then select participants will be scheduled for an in-person screening at the BPRU.

If a participant meets all criteria and agrees to participate, he or she will be enrolled into the study. Enrolled participants will have 2 or 3 sessions involving overnight stays on the Behavioral Pharmacology Research Unit (BPRU) residential unit.

* If participants are on methadone, they will have 2 sessions
* If participants are on buprenorphine, they will have 3 sessions.

Sessions will each last for about 40 hours and involve identical procedures. That means participants will stay 2 nights on the BPRU residential unit for each session, and these sessions will be at least a week a part. Most people will complete all sessions within 1 month.

During sessions participants will experience the following:

Day 1 - Admission to the BPRU residential unit

* Participants will take an alcohol breath test and provide a urine sample to check for drug use (and pregnancy if female). These tests must be negative to be admitted.
* Vital signs will be measured.
* Participants will receive their normal dose of methadone or buprenorphine.

Day 2 - Experimental pain testing

* On each session day, a nurse will insert an IV catheter on the arm or hand not involved with pain testing.
* Investigational drug or placebo will be given in random order. During each pain testing session, participants will receive 4 doses of the same investigational drug or placebo. If participants are on methadone, they will not receive buprenorphine injections as these could cause opioid withdrawal symptoms. Participants will not be told which drug or placebo they are getting and the research staff will not know the assignment either.
* Participants will have 7 rounds of experimental pain testing, each lasting about 45 minutes and consisting of the same pain procedures. A trained technician will show participants each of the pain testing procedures and practice with them until participants learn what is involved and how to respond. Participants will be asked to complete 4 different types of standard pain tests during each session. Participants may stop these procedures at any point by telling the technician that they wish to stop.

  1. One type of test will produce pain by a device that will be pressed against the skin on the shoulder and arm. This produces pressure, similar to pressing a finger against the skin. Participants will be asked to indicate when the pain from the pressure reaches certain levels of intensity.
  2. Another type of test will produce pain by a small device that gives off heat. An investigator will put this device on a participant's forearm and it will increase in temperature. Some of these temperatures will cause participants to experience pain, and they will be asked to rate the pain produced by different intensities of heat.
  3. The third type of pain test will involve placing a hand in very cold water and leaving it there for as long as possible, or until reaching a time limit. Participants will be asked to rate the pain that they feel from the cold water and they may remove their hand from the water at any time.
  4. In addition to pain tests, investigators will also test the ability to detect touch, warmth, and cold sensations. To test for touch sensitivity, a series of very fine threads or thread-like objects will be applied to the forearm and investigators will ask participants to communicate when first noticing any sensation. To test for warmth and cold sensitivity, the same device used to test heat pain sensitivity will be placed on the arm. Participants will be asked to let the investigator know when they first notice the sensation of warmth or cold.

At times, participants will experience more than one type of pain at the same time.

* Participants will answer questions about their experiences, including questions about how the study drug or placebo makes them feel and about any problems with the study drug or placebo.
* Staff will take a participant's vital signs and take a picture of the eye repeatedly over each session.
* Unless participants experience symptoms of opioid withdrawal (for example - nausea, vomiting, diarrhea or loose stools, body aches, and goosebumps), they will not be given the daily dose of methadone or buprenorphine on pain testing day (Day 2).

Day 3 - Discharge

* Vital signs will be measured and a picture of the eye will be taken.
* Participants will answer questions about their experiences from Day 2, including questions about any lasting drug effects and about any problems with the study drug or placebo.
* Participants will receive their normal dose of methadone or buprenorphine and be discharged from the residential unit.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-55;
2. diagnosis of opioid dependence
3. urine toxicology negative for drugs of abuse but positive for opioid maintenance agent;
4. stable buprenorphine (12-16 mg) or methadone (80-100 mg) dose for the past 30 days;
5. absence of acute/chronic pain;
6. able and willing to perform/tolerate pain procedures;
7. able to communicate in English.

Exclusion Criteria:

1. current illicit substance use at screening or during trial (including cannabis use);
2. current diagnosis of alcohol dependence;
3. acute or chronic pain;
4. medical or psychiatric condition known to influence pain testing;
5. current use of prescribed or over the counter analgesic agents;
6. previous allergic reaction to hydromorphone or buprenorphine;
7. women who are pregnant, lactating or planning to get pregnant during the course of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Cold pressor test. | This will be measured 7 times during each 40-hour session. On average, all sessions will be completed within 4 weeks.
  The participant places a hand up to the wrist in a circulating water bath maintained at approximately 4 degrees Celsius (up to 5 minutes). The time at which pain develops is the threshold. The time a volunteer's hand remains underwater before pain is unbearable is tolerance.

SECONDARY OUTCOMES:
Visual analog scales (VAS) of subjective drug effects. | This will be measured 7 times during each 40-hour session. On average, all sessions will be completed within 4 weeks.
  VAS are single item questions that assessed subjective drug effects at the time of scale completion. Ratings are entered into a computer by the participant positioning an arrow along a 100 mm line marked at either end with "none" (0) and "extremely" (100).

CONTACTS AND LOCATIONS:
Overall Officials: D. Andrew Tompkins, M.D., M.H.S., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States